CLINICAL TRIAL: NCT05290818
Title: Total Versus Robotic Assisted Unicompartmental Knee Replacement (TRAKER) for Medial Compartment Osteoarthritis: Randomised Controlled Trial
Brief Title: Total Versus Robotic Assisted Unicompartmental Knee Replacement
Acronym: TRAKER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AC19080
Record Dates: First submitted 2022-02-16; First posted 2022-03-22 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Osteo Arthritis Knee; Arthritis Knee; Arthropathy of Knee
Keywords: Arthroplasty; Robotic; Knee; Total; Partial; Outcome; MAKO
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Intervention Model Description: Randomised control Trial (1:2 ratio: 53 in the rUKA arm and 106 in the mTKA)
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Manual Total Knee Arthroplasty (Active Comparator): This group will receive a conventional manual Triathlon (Stryker) TKA with a cruciate retaining polyethylene insert. The surgeon will then make bone cuts using a manual jig and a hand held saw to prepare the bone surfaces for the implant. A measured resection technique will be employed with a three degree tibial slope. The surgeon will use a conventional jig alignment technique for intramedullary referencing for the femur and extra medullary referencing for the tibia. Once the implant is in position the knee is then balanced by the "feel" though a range of movement and soft tissue releases will be performed as required to balance the knee in flexion and extension.
  Interventions: Device: Triathlon (Stryker) Total Knee Arthroplasty
- Robotic Assisted Unicompartmental Knee Arthroplasty (Experimental): This group will receive the cemented Restoris MCK (Mako, Stryker) with a highly crossed linked (X3) polyethylene insert through a less invasive to the knee joint. Instead of using a manual jig and a hand held burr will be used to prepare the bone surfaces for the implant, the MAKO robotic arm will be used by the surgeon to cut the bone at the required alignment. The information from the CT scan will be used to create a 3D model of the patient's bony anatomy and will used to plan the positioning of the implant. Once the trackers are in place registration of the knee joint surface is performed. The specified bone cuts are then performed using the robotic arm, aiming to gap balance the knee through a full range of movement.
  Interventions: Device: MAKO™ Partial Knee Arthroplasty

INTERVENTIONS:
Device: MAKO™ Partial Knee Arthroplasty — The robotic-arm will be used to position a partial knee arthroplasty.
  Other Names: Robotic-arm assisted partial knee arthroplasty
  Arms: Robotic Assisted Unicompartmental Knee Arthroplasty
Device: Triathlon (Stryker) Total Knee Arthroplasty — Triathlon (Stryker) TKA with a cruciate retaining polyethylene insert.
  Other Names: Total Knee Replacement
  Arms: Manual Total Knee Arthroplasty

SUMMARY:
The purpose of this research is to compare the functional outcomes of patients with end stage medial compartment OA of the knee undergoing a conventional mTKA to those undergoing rUKA and to assess the associated cost economics of such technology.

DETAILED DESCRIPTION:
Unicompartmental knee arthroplasty (UKA) is an accepted surgical alternative to total knee arthroplasty (TKA) for patients with isolated medial compartmental joint disease with the potential advantages of accelerated recovery, improved functional outcomes and retention of anatomical knee kinematics. However, some surgeons continue to favour TKA over UKA due to a lower revision rate. The higher revision rates associated with UKA are thought to be primarily due to component malpositioning and postoperative limb malalignment.

Robotic-arm assisted (r)UKA offers a greater level of precision of component positioning compared to manual UKA and more recently the survivorship of rUKA has been shown to be greater than manual UKA. Early functional outcomes following robotic UKA appear to be better than those observed after manual TKA. Therefore, the benefits of UKA could potentially be enjoyed by the patient without the increased risk of revision when compared to TKA for those with medical compartment disease.

The primary aim of this study is to compare the early knee specific functional outcome of rUKA with manually performed (m)TKA when performed for patients with medial compartment osteoarthritis of the knee.

A single centre randomised control trial will be carried out powered to the Oxford knee score.

ELIGIBILITY:
Inclusion Criteria:

* Listed for elective primary TKA for end stage medial compartment osteoarthritis
* Intact anterior cruciate ligament
* Full thickness and good quality lateral cartilage
* Correctable intra-articular varus deformity and intact medial collateral ligament
* American Society of Anesthesiologists (ASA) grades 1 and 2
* Male or female, age 50 - 75 at the time of listing for surgery
* Suitable candidate for a cruciate retaining TKA (Triathlon prosthesis) and a UKA

Exclusion Criteria:

* Varus deformity of > 20 degrees
* Fixed flexion of >10 degrees
* Patient is unable to comply with the study protocol (incl. refusal for CT scan) or functional assessments
* Female participants who are pregnant, lactating or planning pregnancy during the course of the study
* Requires patella resurfacing or lateral compartment has significant OA
* Inability to understand the patient information for the study, provide written informed consent or answer study questionnaires for cognitive or language reasons
* Inflammatory disorder e.g. rheumatoid arthritis
* Symptomatic foot, hip or spine pathology
* Prior surgery (other than arthroscopy) or septic arthritis of the knee
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study,

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Estimated)
Dates: Start 2024-08-26 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Oxford knee score | Baseline to 6 months
  Knee specific functional outcome measure. It consists of twelve questions assessed on a Likert scale with values from 0 to 4, to give a summative score. This is measured on a scale from 0 (worst) to 48 (best).

SECONDARY OUTCOMES:
Oxford knee score and Activity and Participation Questionnaire | Baseline to 3, 6 and 12 months
  The Oxford knee score is a knee specific functional outcome measure. It consists of twelve questions assessed on a Likert scale with values from 0 to 4, to give a summative score. This is measured on a scale from 0 (worst) to 48 (best). The additional Activity and Participation Questionnaire is a higher functioning supplementary questionnaire consisting of a further eight questions scored 0 (worst) to 4 (best).
Forgotten Joint Score | Baseline to 3, 6 and 12 months
  Knee specific functional outcome. It uses a five-point Likert response format, consisting of 12 equally weighted questions with the raw score transformed to range from zero (worst) to 100 (best) points.
Patient satisfaction | 3, 6 and 12 months
  Patient satisfaction will be assessed following surgery by asking four questions with a different focus:
  i. "Overall how satisfied are you with the results of your knee replacement surgery?" ii. "How satisfied are you with the results of your knee replacement surgery for improving your ability to do housework or yard work (such as cooking, cleaning, or gardening and raking leaves)?" iii. "How satisfied are you with the results of your knee replacement surgery for improving your ability to do recreational activities (such as taking walks, swimming, bicycling, playing golf, dancing, going out with friends)?" iv. "How satisfied are you with the results of your knee replacement surgery for relieving your pain?" The response to each question will be recorded using a four point Likert scale: very satisfied, somewhat satisfied, somewhat dissatisfied, and very dissatisfied.
EQ-5D-3L | Baseline to 3, 6 and 12 months
  Quality of life will be assessed using the EQ-5D-3L general health questionnaire which evaluates five domains (-5D), which include: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. This is a two page questionnaire that consists of five dimensions, with the responses recorded at three levels (3L) of severity (no problems; some problems or extreme problems). The utility index is on a scale of -0.594 to 1, where 1 represents perfect health and a negative value represents a state perceived as worse than death.
  The second page consists of a standard vertical 20cm visual analogue scale (EQ-5D VAS) which is transformed to a scale of 0 (worst) to 100 (best) measuring current health-related quality of life. Each patient's health state, derived from the EQ-5D, will be measured before and after their surgery to determine the change in their health gain or loss after their knee replacement surgery.
Range of movement | Baseline to 3, 6 and 12 months
  A goniometer will be used to measure range of movement by a blinded researcher prior to surgery (baseline), at discharge (immediately post surgery prior to discharge home) and at review appoints. Three measurements will be recorded for extension and flexion of the knee and an average will be documented.
Cost effectiveness | Baseline to 3, 6 and 12 months, and projected for the patients lifetime
  Cost utility analysis will be undertaken to establish the incremental cost effectiveness ratio (ICER). Each patient's health state, derived from the EQ-5D, will be measured before and after their surgery to determine the change in their health gain or loss after their knee replacement surgery. The health state will then be multiplied by the time spent in that state to derive the QALYs gained or lost. The cost per QALY will then be calculated by dividing the cost of the procedure by the QALYs gained after total knee arthroplasty (intervention). A health service resource use questionnaire will be completed by the patient at the 3, 6 and 12 month research assessment. The questionnaire collects data on primary, secondary and community care and associated with the knee replacement over the previous months. Inpatient and surgical data will be collected on the case report forms (CRF's) and complications will be recorded at each visit.
Knee stability and power | Baseline to 3, 6 and 12 months
  Knee stability (stress testing) and power (power rig) will be measured. A stress will be applied to the knee and the joint space opening will be measured using an ultrasound probe which will be used as a marker of knee stability. The power of the knee joint will be assessed using a standardise power rig Specific assessment of the patient's power output will be evaluated by a Leg Extensor Power Rig (Nottingham, UK), well validated for use with this population group.
Patient expectation pre-operative and fulfilment | Baseline to 3, 6 and 12 months
  The Hospital of Special Surgery Expectation questionnaire is a validated measure of patient pre-operative expectations of surgery. The level of patient expectation is indicated on a 5 point Likert scale as 'very important', 'somewhat important', 'a little important', 'I do not expect this' or 'this does not apply to me'. After surgery patients will complete a similar expectation questionnaire, but are asked whether the same expectations had been fulfilled, which again is assessed on a 5 point Likert scale as: 'greatly', 'a lot', 'a little', 'I did not expect this' or 'this did not apply to me'.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas D Clement, MD, PhD, Principal Investigator — NHS Lothian
Locations (1):
- Nicholas Clement, Edinburgh, Lothian, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual patient data available.

REFERENCES:
- [Background] Robinson PG, Clement ND, Hamilton D, Blyth MJG, Haddad FS, Patton JT. A systematic review of robotic-assisted unicompartmental knee arthroplasty: prosthesis design and type should be reported. Bone Joint J. 2019 Jul;101-B(7):838-847. doi: 10.1302/0301-620X.101B7.BJJ-2018-1317.R1. PMID 31256672
- [Background] Clement ND, Bell A, Simpson P, Macpherson G, Patton JT, Hamilton DF. Robotic-assisted unicompartmental knee arthroplasty has a greater early functional outcome when compared to manual total knee arthroplasty for isolated medial compartment arthritis. Bone Joint Res. 2020 May 16;9(1):15-22. doi: 10.1302/2046-3758.91.BJR-2019-0147.R1. eCollection 2020 Jan. PMID 32435451
- [Background] Clement ND, Deehan DJ, Patton JT. Robot-assisted unicompartmental knee arthroplasty for patients with isolated medial compartment osteoarthritis is cost-effective: a markov decision analysis. Bone Joint J. 2019 Sep;101-B(9):1063-1070. doi: 10.1302/0301-620X.101B9.BJJ-2018-1658.R1. PMID 31474149
- [Derived] Clement ND; TRAKER Research Group; Scott CEH, Macpherson GJ, Simpson PM, Leitch G, Patton JT, Ahmed I, Amin AK, Gaston P, Goudie E, Goudie S, Macdonald DM, Martinson E, Moran M, Wade F. Total versus robotic-assisted unicompartmental knee replacement (TRAKER) for medial compartment osteorthritis: a randomized controlled trial. Bone Jt Open. 2025 Feb 10;6(2):164-177. doi: 10.1302/2633-1462.62.BJO-2024-0155.R1. PMID 39923804
- See also: Home page of Edinburgh Orthopaedics — https://edinburghorthopaedics.org/